CLINICAL TRIAL: NCT03339388
Title: Multi-Center Feasibility Study of Enhanced Lithotripsy System (ELS) in The Treatment of Urinary Stone Disease
Brief Title: Enhanced Lithotripsy System (ELS) in the Treatment of Urinary Stone Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adequate enrollment has been achieved
Sponsor: Avvio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-03
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2021-08

CONDITIONS: Urinary Stone
Keywords: lithotripsy; urinary stone
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Enhanced Lithotripsy System (Experimental): Treatment of urinary stones with the Enhanced Lithotripsy System
  Interventions: Device: Enhanced Lithotripsy System

INTERVENTIONS:
Device: Enhanced Lithotripsy System — Stone treatment with the Enhanced Lithotripsy System

SUMMARY:
This is a single arm, multi-center study to assess the safety and efficacy of a form of extracorporeal lithotripsy, called the Enhanced Lithotripsy System, to treat urinary stones.

DETAILED DESCRIPTION:
This is a single arm, multi-center study to assess the safety and efficacy of a form of extracorporeal lithotripsy, called the Enhanced Lithotripsy System, to treat urinary stones. Subjects will be treated up to 2 times with the Enhanced Lithotripsy System and followed for 90 days after the last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years to ≤ 75 years.
* One urinary stone-apparent on a computed tomography (CT) scan within 14 days prior to study enrollment
* Stone size, as estimated by pre-procedure CT, with all dimensions 15 mm or less.
* Provides written informed consent
* Understands and accepts the study requirements

Exclusion Criteria:

* Age less than 18 years of age or over 75 years of age
* Diagnosis of radiolucent stones
* Diagnosis of stones in the lower pole of kidney
* History of cystinuria
* Urine pH below 5.5
* Current untreated urinary tract infection
* Pregnancy
* Coagulation abnormality or taking prescription anticoagulants. Aspirin usage will be discontinued at least 7 days prior to enrollment at the discretion of the attending physician.
* Mobility issues - unable to comfortably lie still for up to 30 minutes or unable to roll from back to side
* Known hypersensitivity to conductivity gel
* Vulnerable individuals (mentally disabled, physically disabled, prisoner, etc.)
* Body mass index greater than 35
* American Society of Anesthesiologists (ASA) score of 3 or greater general anesthesia risk level
* Known sensitivity to possible medications used before, during, or after the ELS procedure, including but not limited to the following: sedative agents, general anaesthetics, topical anaesthetics, and opioid analgesics.
* Enrollment in another research study or previous participation within 30 days of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Proportion of study participants with Serious Device and/or Serious Procedure-Related Adverse Events (Safety) | 90 days
  Incidence of Serious Device and/or Serious Procedure-Related adverse events

SECONDARY OUTCOMES:
Stone-free status | 30 days
  Proportion of study participants who are successfully treated [absence of stones or with only clinically-insignificant remaining fragments]

OTHER OUTCOMES:
Pain medication usage | 30 days
  Collection of pain concomitant pain medications
Time to stone passage | 30 days
  Evaluation of stone presence
Pain scoring | 30 days
  Patient reported pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Damien M Bolton, MD, MBBS, Principal Investigator — Austin Hospital, Melbourne Australia
Locations (4):
- Australia (4):
  - McArthur Urology, Campbelltown, New South Wales
  - Westmead Private Hospital, Westmead, New South Wales
  - Goldfields Urology, Bendigo, Victoria
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No